CLINICAL TRIAL: NCT01015313
Title: A Multi-center, Randomized, Controlled and Prospective Pilot Study on the Effects of Intensified Sodium Management on Hospitalization in Chronic Hemodialysis Patients.
Brief Title: Effects of Intensified Sodium Management in Hemodialysis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 208-12 (formerly 173-09)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: sodium, hypertension, volume overload
MeSH Terms: conditions — Hypertension; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive sodium management (Experimental)
  Interventions: Other: intensive sodium management
- standard care (No Intervention)

INTERVENTIONS:
Other: intensive sodium management — 1. dietary sodium restriction
  2. avoiding positive sodium balance during dialysis by: aligning dialysate sodium with plasma sodium, avoiding sodium profiling, and avoiding saline solutions to treat intradialytic symptoms
  Arms: intensive sodium management

SUMMARY:
The primary aim of this study is to investigate whether intensive sodium management by dietary sodium restriction and by preventing positive sodium balance during dialysis can be successfully applied in chronic hemodialysis patients. Secondary aims are to test if sodium restriction has positive effects on the frequency of hospital admissions, blood pressure, fluid overload, quality of life and residual renal function.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, clinically stable maintenance hemodialysis patients on a thrice weekly HD regimen.
* Willing and able to provide written, signed informed consent after the nature of the study has been explained.
* Willing and able to comply with all study procedures.
* Age ≥18 years.

Exclusion Criteria:

* Simultaneous participation in another clinical study except observational trials.
* Any psychological condition which could interfere with the patient's ability to comply with the study protocol.
* Pregnancy.
* Amputation of a limb.
* Pacemaker, implantable pump, artificial joint.
* Expectation that native kidney function will recover.
* Unable to verbally communicate in English or Spanish.
* Scheduled for living donor kidney transplant, change to peritoneal dialysis, home HD or plans to relocate to another center within the next 14 months.
* Life expectancy < 15 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
feasibility of intensive sodium management | 12 months

SECONDARY OUTCOMES:
hospitalization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute; Nathan W Levin, MD, Study Director — Renal Research Institute
Locations (3):
- United States (3):
  - Irving Place Dialysis Center, New York, New York
  - Upper Manhattan Dilaysis Center, New York, New York
  - Yorkville Dialysis Center, New York, New York

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803